CLINICAL TRIAL: NCT02573428
Title: Evaluating the Validity of an Eye Gaze Tracking Assessment Tool in Identifying Autism Spectrum Disorder
Brief Title: Evaluating the Validity of an Eye Gaze Paradigm in Predicting Autism Spectrum Disorder
Acronym: EYE
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Thomas W. Frazier, Ph.D, Director, Center for Autism, The Cleveland Clinic
Other Study IDs: 14-620
Record Dates: First submitted 2015-10-07; First posted 2015-10-09 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Autism Spectrum Disorders
Keywords: Autism Spectrum Disorder; Eye Gaze; Remote Eye Gaze Tracking; Autism
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Autism Spectrum Disorder: Individuals who receive a clinical diagnosis of Autism Spectrum Disorder
- Developmental/Psychiatric Controls: Individuals who receive a clinical diagnosis of another developmental or psychiatric disorder
- Healthy Controls: Individuals who have no specific developmental or psychiatric diagnosis

SUMMARY:
The primary purpose of the present study is to evaluate the diagnostic validity of eye tracking measurements acquired during viewing of socially-relevant stimuli in predicting ASD diagnosis. The secondary purpose was to explore the potential prognostic value of eye tracking measures through cross-sectional associations with non-verbal cognitive ability.

Deficits in eye gaze are a hallmark sign of autism. A large and growing body of research supports the ability of eye-tracking based measurements to sensitively discriminate individuals with ASD and healthy participants. These investigations have identified that the core deficit in autism as disruption of social attention, reflecting an inability to appropriately engage and track socially- and emotionally-relevant aspects of the visual world. Thus, eye gaze tracking, acquired during viewing of socially-relevant stimuli, may be a useful approach to identifying objective markers of ASD. Eye tracking also carries the advantages of being less intrusive and expensive than MRI and genetic testing and specifically focuses on the core neurobehavioral characteristics of ASD - abnormalities in social attention.

After diagnosis of ASD, key clinical tasks in young children involve determining an accurate prognosis and tracking the progress of early interventions. Currently, the only prognostic indicators are clinical observations (subjective and expensive) and non-verbal cognitive ability testing (difficult to acquire, time-consuming, unavailable in many settings). Recently, eye gaze tracking was found to predict functional outcomes. Thus, in addition to being an objective marker for ASD, eye tracking measurements have potential to be useful for predicting cognitive and functional outcomes. Similarly, the only available methods for tracking treatment progress are parental reports (highly subjective), clinical observations (subjective and expensive), and cognitive measurements (expensive and unavailable in many settings. This study will evaluate, using cross-section data, the potential for eye tracking data to serve as a proxy for non-verbal cognitive ability scores in determining prognosis for ASD-affected children. Additionally, this study will evaluate the test re-test reliability of eye tracking parameters that can potentially be used to track treatment progress.

DETAILED DESCRIPTION:
The current study will occur in four phases: pilot testing, development, validation, and re-test. In each phase, participants will view a visual attention stimulus with social elements (social attention paradigm) while eye tracking measurements are remotely acquired. The visual attention paradigm will be refined in the pilot testing but will remain the same for development, validation, and re-test phases. The entire process, including calibration and viewing of the visual paradigm, will take about 15 minutes. The text below describes each phase in detail and the reviews specific methodology for the social attention paradigm and eye tracking procedures.

1. Pilot Phase. Pilot testing of the social attention paradigm used to elicit eye gaze measurements to ensure they are sufficiently engaging across the ages of children participating. The visual attention paradigm during this phase is expected to be 10-12 minutes. This phase will also be used to determine optimal strategies for maintaining attention throughout the testing period. Initial data may also provide some insights into the most discriminating stimulus elements to include in future phases. Investigators anticipate recruiting approximately 10 ASD and 10 non-ASD participants in this phase. The pilot phase is expected to require 2.5 months of recruitment and 0.5 months of data reduction and analysis.
2. Development Phase. Once pilot testing is completed, 30 ASD-affected and 30 non-ASD children ages 1.5 to 18 will be recruited. Each child will complete the social attention paradigm while their eye gaze is remotely tracked. Eye gaze data is then scored for more than 100 parameters and these scores are entered into a database that includes diagnostic and cognitive information about each participant. The eye tracking data is then analyzed to create the diagnostic and prognostic algorithms that will refine the system's diagnostic sensitivity and specificity in the ASD population. The development period will require 6 months of data collection, followed by 3 months of scoring and algorithm computation.
3. Validation Phase. Collection of the validation sample will include 60 ASD-affected and 60 non-ASD affected children ages 1.5-18. The validation phase will use the same visual social attention paradigm and methods used in the development sample. The validation period will overlap algorithm development and require 8 months of data collection and 1 month of analysis.
4. Re-Test Phase. Participants in the re-test phase will include 30 ASD and 30 non-ASD children recruited in the first half of the validation phase. These participants will be explained in the validation phase that investigators will be re-recruiting them for the re-test phase approximately 3-6 months following their initial testing during the validation phase.

The target sample size varies depending on the phase of the study. Below are the target sample sizes for each phase:

Pilot Phase = 10 ASD and 10 Non-ASD Development Phase = 30 ASD and 30 Non-ASD Validation Phase = 60 ASD and 60 Non-ASD Re-Test Phase = 30 ASD and 30 Non-ASD (from the validation phase) The study population is individuals with autism spectrum disorder, or a clinical diagnosis of another developmental or psychiatric disorder (developmental/psychiatric controls), or have no specific developmental or psychiatric diagnosis (healthy controls), ages 1.5 (18 months) to 18 (120 months) at time of consent.

Eye gaze data will be collected using a remote eye tracker from Sensori-motoric instruments (SMI). Remote eye tracking offers minimal invasiveness to the viewer's field of view and collects time-stamped, 3D eye position, and binocular gaze and pupil data at a sampling rate of 120 Hz. Eye gaze capture is automatically calibrated to 2/5/9 points and provides position accuracy to 0.5° at a 60cm viewing distance. Gaze tracking data, screen recordings, user events, and gaze position will be recorded simultaneously. Data will be analyzed with emphasis on areas-of- interest and dwell time on specific targets on a second-by-second basis. Examples of the types of measures captured include: dwell time to any area of the stimulus, dwell time to the face and non-face regions of a human form on the video, fixation shifts between stimuli.

Additional tests and demographic data will be collected from standard of care autism diagnostic and behavioral health diagnostic appointments that can be found in the medical record.

Pilot Analyses. In the pilot phase, investigators will compute the effect size (Cohen's d) between ASD and non-ASD participants for each of the eye gaze parameters acquired for each of the individual stimuli in the social attention paradigm. Stimulus elements eliciting the largest discrimination between ASD and non-ASD patients will be retained in the development phase.

ASD Diagnostic Algorithm Analyses. In the development phase, all of the eye gaze measurements acquired from the social attention paradigm will be included as predictor variables in a random forest analysis. This analysis permits evaluation of the discriminative ability of a large number of variables in data sets with a modest number of cases. The variables with highest importance scores, indicating good diagnostic discrimination, will be entered into a logistic regression analysis with ASD diagnostic status (ASD vs. non-ASD) as the dichotomous dependent variable. Significant predictors will be retained and coefficients from the retained predictors will serve as the diagnostic algorithm.

The diagnostic algorithm scores will then be submitted to Receiver Operating Characteristic (ROC) curve analyses to provide detailed evaluation of sensitivity and specificity of the algorithm in the detection of ASD. Areas under the curve of >.90 are expected, indicating strong diagnostic validity.

Prognostic Algorithm Analyses. To identify a prognostic algorithm, a similar process will be conducted with all the available eye tracking measurements as predictors and non-verbal cognitive ability scores (dichotomized at <70 and 70 and above) as the dependent variable in random forest analyses. Non-verbal cognitive ability scores will be dichotomized based on previous data suggesting that individuals with ASD and intellectual disability show worse outcome. The predictor variables with highest importance, indicating good diagnostic discrimination, will then be entered into a logistic regression analysis with non-verbal cognitive ability (<70, >=70) as the dichotomous dependent variable. Significant predictors will be retained and coefficients from the retained predictors will serve as the prognostic algorithm. The prognostic algorithm scores will then be submitted to Receiver Operating Characteristic (ROC) curve analyses to provide detailed evaluation of sensitivity and specificity of the algorithm in the detection of non-verbal cognitive disability. Areas under the curve of >.80 are expected, indicating good validity in predicting cognitive disability. Non-verbal cognitive ability will be the primary focus of these analyses because of its documented relationship with outcome in individuals with autism. However, similar analyses will be computed for verbal cognitive ability and adaptive function scores. Investigators will also conduct the above analyses using continuous measurements as dichotomization may unnecessarily deflate validity.

Treatment Tracking Algorithm Analyses. To identify a treatment tracking algorithm, investigators will simply combine the eye tracking measurements identified in the diagnostic and prognostic algorithm into a single treatment tracking algorithm. To evaluate test re-test reliability of these measurements investigators will use intra-class correlation coefficients (model 2 - absolute agreement).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Autism Spectrum Disorder (299.0) following evaluation in Cleveland Clinic Center for Autism Diagnostic Clinic, or a clinical diagnosis of another developmental or psychiatric disorder, or have no specific developmental or psychiatric diagnosis.
* Age 1.5 to 18 years at time of consent.

Exclusion Criteria:

* Individuals whom, with corrective lenses are still legally blind.
* Individuals whom, it is determined at the discretion of hte Primary Investigator, after consultation with the evaluating psychologist in the Center for Autism Diagnostic Clinic, are not able to sufficiently attend to the stimulus presentation or have substantial challenging behaviors that would prohibit participation.

Ages: 18 Months to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: ASD and Non-ASD participants will be recruited following their evaluations in the Center for Autism diagnostic clinics as well as from the Social Practice and Instruction Enhances Socialization (SPIES) program both of which are part of the Cleveland Clinic Center for Autism.
Sampling Method: Non-Probability Sample
Enrollment: 389 (Actual)
Dates: Start 2015-06; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Percentage of correctly discriminated ASD and non-ASD cases using the autism risk index. | 1 year from study start
  In the development phase, all of the eye gaze measurements acquired from the social attention paradigm will be included as predictor variables in a random forest analysis. This analysis permits evaluation of the discriminative ability of a large number of variables in data sets with a modest number of cases. The variables with highest importance scores, indicating good diagnostic discrimination, will be entered into a logistic regression analysis with ASD diagnostic status (ASD vs. non-ASD) as the dichotomous dependent variable. Significant predictors will be retained and coefficients from the retained predictors will serve as the diagnostic autism risk index.

SECONDARY OUTCOMES:
Area under the ROC curve of the prognostic algorithm in discriminating non-verbal cognitive disability. | 21 months from study start
  All the available eye tracking measurements as predictors and non-verbal cognitive ability scores (dichotomized at <70 and 70 and above) as the dependent variable in random forest analyses.
Number of regions of interest with significant dwell time differences between ASD-affected and non-ASD participants. | 3 months from study start
  Effect size between ASD and non-ASD participants for dwell time relative to social targets presented in the social attention paradigm.
Natural Interaction, Monologue with Directed Attention Stimulus - Dwell time in Upper Face Region of Interest (ROI) from 0.5-24 seconds | 6 months from study start
Natural Interaction, Monologue with Directed Attention Stimulus - Dwell time in Desk picture and Cup/Phone Regions of Interest (ROI) from 0.5-24 seconds | 6 months from study start
Natural Interaction, Joke 1 Stimulus - Dwell time in the Upper and Lower Face ROIs from 0.5-5.5 seconds | 6 months from study start
Natural Interaction, Joke 1 Stimulus - Dwell time in Body and Toys ROIs from 0.5-6.88 seconds | 6 months from study start
Natural Interaction, Joke 2 Stimulus - Dwell time in Upper Face ROI and Lower Face ROI from 0.5-8.0 seconds | 6 months from study start
Natural Interaction, Joke 2 Stimulus - Dwell time in Upper Face ROI from 4.3-5.0 seconds | 6 months from study start
Natural Interaction, Joke 2 Stimulus - Dwell time in Distractor 1, Distractor 2, Distractor 3 and Body ROIs from 0.2-10.34 seconds | 6 months from study start
Joint Attention, Gaze Middle Stimulus - Dwell time in Face ROI from 0.3-1.1 seconds | 6 months from study start
Joint Attention, Gaze Middle Stimulus - Dwell time in Target Toy, Distractor Right and Distractor Left ROIs from 1.0-2.3 seconds | 6 months from study start
Joint Attention, Gaze Right Stimulus - Dwell time in Face A and Face B ROIs from 3.3-3.7 seconds | 6 months from study start
Joint Attention, Gaze Right Stimulus - Dwell time in Target Toy and Distractor Toy ROIs from 1.0-2.3 seconds | 6 months from study start
Joint Attention, Gaze Right 2 Stimulus - Dwell time in Face ROI from 2.0-3.0 | 6 months from study start
Joint Attention, Gaze Right 2 Stimulus - Dwell time in Left Distractor, Middle Distractor and Right Target from 0.9-1.6 seconds | 6 months from study start
Joint Attention, Gesture Middle 1 Stimulus - Left Distractor, Right Distractor and Middle Target from 1.5-3.5 seconds | 6 months from study start
Joint Attention, Gesture Right 1 Stimulus - Target Toy, Distractor Middle and Distractor Left ROIs from 0.8-3.5 seconds | 6 months from study start
Joint Attention, Gesture Right 2 Stimulus - Target Toy and Distractor Toy ROIs from 1.3-2.4 seconds | 6 months from study start
Joint Attention, Gesture Left 1 Stimulus - Target Toy, Distractor Middle and Distractor Right ROIs from 1.4-3.4 seconds | 6 months from study start
Joint Attention, Gesture Left 2 Stimulus - Target Toy and Distractor Right ROIs from 1.2-2.7 seconds | 6 months from study start
Joint Attention - Gesture Left 3 Stimulus - Left Target, Middle Distractor and Right Distractor ROIs from 0.7-2.3 seconds | 6 months from study start

OTHER OUTCOMES:
Natural Interaction, Monologue with Directed Attention Stimulus - Dwell time in Face Region of Interest (ROI) from 0.5-8.0 seconds. | 6 months from study start
Natural Interaction, Monologue with Directed Attention Stimulus - Dwell time in Cup/Phone, Desk Picture, Wall Picture and Light Switch ROIs from 0.2-24.0 seconds | 6 months from study start
Side by Side Faces, Male Sad Target Stimulus - Dwell time in Target Upper Face ROI from 0.3-0.5 seconds | 6 months from study start
Side by Side Faces, Male Sad Target Stimulus - Dwell time in Distracter Face ROI from 0.7-1.1 seconds | 6 months from study start
Side by Side Faces, Male Sad Target Stimulus - Dwell time in Target Upper Face ROI from 1.5-5.0 seconds | 6 months from study start
Side by Side Faces, Male Sad Target Stimulus - Dwell time in Distrater Face, Target Body, and Distracter Body ROI from 1.5-5.0 seconds | 6 months from study start
Side by Side Faces, Female Scared Target Stimulus - Dwell time Target Upper Face ROI from 0.5-0.8 seconds | 6 months from study start
Side by Side Faces, Female Scared Target Stimulus - Dwell time Target Upper Face ROI from 1.9-5.0 seconds | 6 months from study start
Side by Side Faces, Female Scared Target Stimulus - Dwell time Distracter Face, Target Body, and Distracter Body ROI from 1.9-5.0 seconds | 6 months from study start
Side by Side Faces, Female Surpised Target Stimulus - Dwell time Target Upper Face ROI from 1.8-5.0 seconds | 6 months from study start
Side by Side Faces, Female Surpised Target Stimulus - Dwell time Distracter Face, Target Body, and Distracter Body ROI from 1.8-5.0 seconds | 6 months from study start
Side by Side Faces, Female Sad Target Stimulus - Dwell time Target Upper Face ROI from 1.3-5.0 seconds | 6 months from study start
Side by Side Faces, Female Sad Target Stimulus - Dwell time Distracter Face, Target Body,and Distracter Body ROI from 1.3-5.0 seconds | 6 months from study start
Side by Side Faces, Male Happy Target Stimulus - Dwell time Target Upper Face ROI from 2.0-5.0 seconds | 6 months from study start
Side by Side Faces, Male Happy Target Stimulus - Dwell time Distracter Face, Target Body, and Distracter Face ROI from 2.0-5.0 seconds | 6 months from study start
Side by Side Faces, Male Angry Target Stimulus - Dwell time Target Upper Face ROI from 1.7-5.0 seconds | 6 months from study start
Side by Side Faces, Male Angry Target Stimulus - Dwell time Target Lower Face ROI from 1.7-5.0 seconds | 6 months from study start
Side by Side Faces, Male Angry Target Stimulus - Dwell time Distracter Face, Target Body, and Distracter Body ROI from 1.7-5.0 seconds | 6 months from study start
Face vs. Abstract Design 1 Stimulus - Dwell time Upper Face ROI from 0.5-10.0 seconds | 6 months from study start
Face vs. Abstract Design 1 Stimulus - Dwell time Abstract ROI from 0.5-10.0 seconds | 6 months from study start
Biological vs. Non-Biological Motion, Scramble vs. Give Me Stimulus - Dwell time Predictive Action ROI from 1.1 to 1.5 seconds | 6 months from study start
Biological vs. Non-Biological Motion, Scramble vs. Give Me Stimulus - Dwell time Predictive Action ROI from 3.4 to 4.3 seconds | 6 months from study start
Joint Attention, Gaze Middle 1 Stimulus - Dwell time Face ROI from 0.4 to 1.0 seconds | 6 months from study start
Joint Attention, Gaze Middle 1 Stimulus - Dwell time Target Toy ROI from 1.0 to 2.3 seconds | 6 months from study start
Joint Attention, Gaze Middle 1 Stimulus - Dwell time Distracter Right, and Distracter Left ROI from 1.0 to 2.3 seconds | 6 months from study start
Joint Attention, Gaze Middle 1 Stimulus - Dwell time Face ROI from 2.4 to 3.0 seconds | 6 months from study start
Joint Attention, Gesture Right 1 Stimulus - Dwell time Face ROI from 2.0 to 3.5 seconds | 6 months from study start
Joint Attention, Gesture Right 1 Stimulus - Dwell time Gesture ROI from 0.6 to 3.3 seconds | 6 months from study start
Joint Attention, Gesture Right 1 Stimulus - Dwell time Target Toy ROI from 0.8 to 2.8 seconds | 6 months from study start
Joint Attention, Gesture Right 1 Stimulus - Dwell time Distracter Middle, and Distracter Left ROI from 0.8 to 2.8 seconds | 6 months from study start
Joint Attention, Gesture Left 1 Stimulus - Dwell time Face ROI from 0.3 to 1.0 seconds | 6 months from study start
Joint Attention, Gesture Left 1 Stimulus - Dwell time Gesture ROI from 1.1 to 3.2 seconds | 6 months from study start
Joint Attention, Gesture Left 1 Stimulus - Dwell time Target Toy ROI from 1.4 to 3.4 seconds | 6 months from study start
Joint Attention, Gesture Left 1 Stimulus - Dwell time Distracter Right, and Distracter Middle ROI from 1.4 to 3.4 seconds | 6 months from study start
Face vs. Abstract Design 2 Stimulus - Dwell time Upper Face ROI from 0.7 to 10.0 seconds | 6 months from study start
Face vs. Abstract Design 2 Stimulus - Dwell time Abstract ROI from 0.7 to 10.0 seconds | 6 months from study start
Biological vs. Non-Biological Motion, Scramble vs. Which One Stimulus - Dwell time Predictive Action ROI from 1.3 to 5.0 seconds | 6 months from study start
Biological vs. Non-Biological Motion, Scramble vs. Help Self Stimulus - Dwell time Predictive Action ROI from 4.9 to 5.5 seconds | 6 months from study start
Natural Interaction, Gesture Stop Stimulus - Dwell time Female Face ROI from 0.5 to 18.28 seconds | 6 months from study start
Natural Interaction, Gesture Stop Stimulus - Dwell time Male Face ROI from 0.5 to 18.28 seconds | 6 months from study start
Natural Interaction, Gesture Stop Stimulus - Dwell time Bubble Wrap ROI from 4.1 to 5.4 seconds | 6 months from study start
Natural Interaction, Gesture Stop Stimulus - Dwell time Bubble Wrap ROI from 10.0 to 11.5 seconds | 6 months from study start
Natural Interaction, Gesture Stop Stimulus - Dwell time Monitor, Laptop, Desk Picture, and Pencil Cup ROI from 0.2 to 18.28 seconds | 6 months from study start
Natural Interaction, Reciprocal Conversation Stimulus - Dwell time Female Face ROI from 0.5 to 16.34 seconds | 6 months from study start
Natural Interaction, Reciprocal Conversation Stimulus - Dwell time Male Face ROI from 0.5 to 16.34 seconds | 6 months from study start
Natural Interaction, Reciprocal Conversation Stimulus - Dwell time Hats ROI from 1.5 to 3.5 seconds | 6 months from study start
Natural Interaction, Reciprocal Conversation Stimulus - Dwell time Hats ROI from 9.5 to 16.34 seconds | 6 months from study start
Natural Interaction, Drink Spill Stimulus - Dwell time Face 1 ROI from 2.4 to 2.9 seconds | 6 months from study start
Natural Interaction, Drink Spill Stimulus - Dwell time Face 2 ROI from 3.2 to 3.7 seconds | 6 months from study start
Natural Interaction, Drink Spill Stimulus - Dwell time Pitcher/Glass Spill ROI from 4.3 to 8.6 seconds | 6 months from study start
Natural Interaction, Drink Spill Stimulus - Dwell time Face 1 Expression ROI from 9.0 to 11.88 seconds | 6 months from study start
Natural Interaction, Drink Spill Stimulus - Dwell time Face 2 ROI from 10.0 to 11.88 seconds | 6 months from study start
Natural Interaction, Joke 1 Stimulus - Dwell time Upper Face ROI from 0.5 to 6.88 seconds | 6 months from study start
Natural Interaction, Joke 1 Stimulus - Dwell time Body, and Toys ROI from 0.5 to 6.88 seconds | 6 months from study start
Natural Interaction, Tap Shoulder Stimulus - Dwell time Male Face ROI from 0.3 to 12.29 seconds | 6 months from study start
Natural Interaction, Tap Shoulder Stimulus - Dwell time Female Face ROI from 2.2 to 12.29 seconds | 6 months from study start
Natural Interaction, Tap Shoulder Stimulus - Dwell time Tap ROI from 6.4 to 7.1 seconds | 6 months from study start
Natural Interaction, Tap Shoulder Stimulus - Dwell time Paper ROI from 0.2 to 12.29 seconds | 6 months from study start
Natural Interaction, Offer to Share Stimulus - Dwell time Face A ROI from 0.6 to 3.2 seconds | 6 months from study start
Natural Interaction, Offer to Share Stimulus - Dwell time Face B and Gesture/Shrug ROI from 3.8 to 6.7 seconds | 6 months from study start
Natural Interaction, Offer to Share Stimulus - Dwell time Face A ROI from 7.2 to 9.1 seconds | 6 months from study start
Natural Interaction, Offer to Share Stimulus - Dwell time Orange/Hands ROI from 9.4 to 11.3 seconds | 6 months from study start
Dynamic Facial Expression, Happy Stimulus - Dwell time Upper Face ROI from 0.2 to 4.0 seconds | 6 months from study start
Dynamic Facial Expression, Angry Stimulus - Dwell time Upper Face ROI from 0.2 to 0.8 seconds | 6 months from study start
Dynamic Facial Expression, Angry Stimulus - Dwell time Lower Face ROI from 0.9 to 1.2 seconds | 6 months from study start
Dynamic Facial Expression, Angry Stimulus - Dwell time Upper Face ROI from 1.3 to 2.2 seconds | 6 months from study start
Dynamic Facial Expression, Sad Stimulus - Dwell time Upper Face ROI from 0.6 to 4.0 seconds | 6 months from study start
Dynamic Facial Expression, Surprise Stimulus - Dwell time Upper Face ROI from 0.5 to 1.6 seconds | 6 months from study start
Joint Attention, Gesture Left 2 Stimulus - Dwell time Face B ROI from 0.7 to 1.1 seconds | 6 months from study start
Joint Attention, Gesture Left 2 Stimulus - Dwell time Target ROI from 1.2 to 2.7 seconds | 6 months from study start
Joint Attention, Gesture Left 2 Stimulus - Dwell time Distracter Right ROI from 1.2 to 2.7 seconds | 6 months from study start
Joint Attention, Gesture Left 2 Stimulus - Dwell time Face A ROI from 1.4 to 3.2 seconds | 6 months from study start
Joint Attention, Gaze Right Stimulus - Dwell time Face B-male ROI from 0.7 to 2.5 seconds | 6 months from study start
Joint Attention, Gaze Right Stimulus - Dwell time Face B-male ROI from 3.1 to 3.7 seconds | 6 months from study start
Joint Attention, Gesture Right 2 Stimulus - Dwell time Face B ROI from 0.8 to 1.1 seconds | 6 months from study start
Joint Attention, Gesture Right 2 Stimulus - Dwell time Face B ROI from 2.6 to 3.2 seconds | 6 months from study start
Joint Attention, Gesture Right 2 Stimulus - Dwell time Target & Gesture ROI from 1.0 to 2.0 seconds | 6 months from study start
Joint Attention, Gesture Right 2 Stimulus - Dwell time Distracter ROI from 1.0 to 2.0 seconds | 6 months from study start
Dynamic Facial Expressions, Surprise 2 Stimulus - Dwell time Upper Face ROI from 0.4 to 1.3 seconds | 6 months from study start
Dynamic Facial Expressions, Surprise 2 Stimulus - Dwell time Lower Face ROI from 1.5 to 1.7 seconds | 6 months from study start
Dynamic Facial Expressions, Surprise 2 Stimulus - Dwell time Upper Face ROI from 1.8 to 4.0 seconds | 6 months from study start
Dynamic Facial Expressions, Angry 2 Stimulus - Dwell time Upper Face ROI from 0.3 to 1.8 seconds | 6 months from study start
Dynamic Facial Expressions, Angry 2 Stimulus - Dwell time Upper Face ROI from 2.5 to 4.0 seconds | 6 months from study start
Dynamic Facial Expressions, Happy 2 Stimulus - Dwell time Upper Face ROI from 2.5 to 4.0 seconds | 6 months from study start
Dynamic Facial Expressions, Scared Stimulus - Dwell time Upper Face ROI from 3.5 to 3.8 seconds | 6 months from study start
Natural Interaction, Joke 2 Stimulus - Dwell time Upper Face ROI from 2.0 to 8.0 seconds | 6 months from study start
Natural Interaction, Joke 2 Stimulus - Dwell time Distracter 1, Distracter 2, Distracter 3, and Microphone ROI from 0.2 to 10.34 seconds | 6 months from study start
Joint Attention, Gaze Right 2 Stimulus - Dwell time Face ROI from 0.5 to 0.8 seconds | 6 months from study start
Joint Attention, Gaze Right 2 Stimulus - Dwell time Left Distracter, and Middle Distracter ROI from 0.9 to 1.6 seconds | 6 months from study start
Joint Attention, Gaze Right 2 Stimulus - Dwell time Right Target ROI from 0.9 to 1.6 seconds | 6 months from study start
Joint Attention, Gesture Middle Stimulus - Dwell time Face ROI from 0.4 to 0.6 seconds | 6 months from study start
Joint Attention, Gesture Middle Stimulus - Dwell time Left Distracter, and Right Distracter ROI from 1.5 to 3.0 seconds | 6 months from study start
Joint Attention, Gesture Middle Stimulus - Dwell time Gesture and Middle Target ROI from 1.5 to 3.0 seconds | 6 months from study start
Joint Attention, Gesture Middle Stimulus - Dwell time Face ROI from 3.4 to 4.0 seconds | 6 months from study start
Joint Attention, Gesture Left 3 Stimulus - Dwell time Face ROI from 0.3 to 0.5 seconds | 6 months from study start
Joint Attention, Gesture Left 3 Stimulus - Dwell time Left Target, Middle Distracter, and Right Distracter ROI from 0.7 to 2.3 seconds | 6 months from study start
Joint Attention, Gesture Left 3 Stimulus - Dwell time Gesture ROI from 0.8 to 1.8 seconds | 6 months from study start

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Frazier, Ph.D., Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Center for Autism, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ritvo ER, Freeman BJ, Pingree C, Mason-Brothers A, Jorde L, Jenson WR, McMahon WM, Petersen PB, Mo A, Ritvo A. The UCLA-University of Utah epidemiologic survey of autism: prevalence. Am J Psychiatry. 1989 Feb;146(2):194-9. doi: 10.1176/ajp.146.2.194. PMID 2783539
- [Background] Fombonne E. Epidemiology of autistic disorder and other pervasive developmental disorders. J Clin Psychiatry. 2005;66 Suppl 10:3-8. PMID 16401144
- [Background] Developmental Disabilities Monitoring Network Surveillance Year 2010 Principal Investigators; Centers for Disease Control and Prevention (CDC). Prevalence of autism spectrum disorder among children aged 8 years - autism and developmental disabilities monitoring network, 11 sites, United States, 2010. MMWR Surveill Summ. 2014 Mar 28;63(2):1-21. PMID 24670961
- [Background] Ganz ML. The costs of autism. In: Moldin SO, Rubenstein JLR, eds. Understanding autism: From basic neuroscience to treatment: CRC Press; 2006.
- [Background] Ganz ML. The lifetime distribution of the incremental societal costs of autism. Arch Pediatr Adolesc Med. 2007 Apr;161(4):343-9. doi: 10.1001/archpedi.161.4.343. PMID 17404130
- [Background] Pierce K, Carter C, Weinfeld M, Desmond J, Hazin R, Bjork R, Gallagher N. Detecting, studying, and treating autism early: the one-year well-baby check-up approach. J Pediatr. 2011 Sep;159(3):458-465.e1-6. doi: 10.1016/j.jpeds.2011.02.036. Epub 2011 Apr 27. PMID 21524759
- [Background] Ozonoff S, Iosif AM, Baguio F, Cook IC, Hill MM, Hutman T, Rogers SJ, Rozga A, Sangha S, Sigman M, Steinfeld MB, Young GS. A prospective study of the emergence of early behavioral signs of autism. J Am Acad Child Adolesc Psychiatry. 2010 Mar;49(3):256-66.e1-2. PMID 20410715
- [Background] Grice SJ, Halit H, Farroni T, Baron-Cohen S, Bolton P, Johnson MH. Neural correlates of eye-gaze detection in young children with autism. Cortex. 2005 Jun;41(3):342-53. doi: 10.1016/s0010-9452(08)70271-5. PMID 15871599
- [Background] Lord, RM, DiLavore PC, et al. Autism Diagnostic Observation Schedule: WPS (ADOS-WPS). Los Angeles, CA: Western Psychological Services. 1999.
- [Background] Volkmar FR, Lord C, Bailey A, Schultz RT, Klin A. Autism and pervasive developmental disorders. J Child Psychol Psychiatry. 2004 Jan;45(1):135-70. doi: 10.1046/j.0021-9630.2003.00317.x. PMID 14959806
- [Background] Bolton PF, Golding J, Emond A, Steer CD. Autism spectrum disorder and autistic traits in the Avon Longitudinal Study of Parents and Children: precursors and early signs. J Am Acad Child Adolesc Psychiatry. 2012 Mar;51(3):249-260.e25. doi: 10.1016/j.jaac.2011.12.009. Epub 2012 Feb 3. PMID 22365461
- [Background] Kozlowski AM, Matson JL, Horovitz M, Worley JA, Neal D. Parents' first concerns of their child's development in toddlers with autism spectrum disorders. Dev Neurorehabil. 2011;14(2):72-8. doi: 10.3109/17518423.2010.539193. PMID 21410398
- [Background] Jones W, Klin A. Attention to eyes is present but in decline in 2-6-month-old infants later diagnosed with autism. Nature. 2013 Dec 19;504(7480):427-31. doi: 10.1038/nature12715. Epub 2013 Nov 6. PMID 24196715
- [Background] Chawarska K, Macari S, Shic F. Decreased spontaneous attention to social scenes in 6-month-old infants later diagnosed with autism spectrum disorders. Biol Psychiatry. 2013 Aug 1;74(3):195-203. doi: 10.1016/j.biopsych.2012.11.022. Epub 2013 Jan 11. PMID 23313640
- [Background] Wolff JJ, Gu H, Gerig G, Elison JT, Styner M, Gouttard S, Botteron KN, Dager SR, Dawson G, Estes AM, Evans AC, Hazlett HC, Kostopoulos P, McKinstry RC, Paterson SJ, Schultz RT, Zwaigenbaum L, Piven J; IBIS Network. Differences in white matter fiber tract development present from 6 to 24 months in infants with autism. Am J Psychiatry. 2012 Jun;169(6):589-600. doi: 10.1176/appi.ajp.2011.11091447. PMID 22362397
- [Background] Chawarska K, Campbell D, Chen L, Shic F, Klin A, Chang J. Early generalized overgrowth in boys with autism. Arch Gen Psychiatry. 2011 Oct;68(10):1021-31. doi: 10.1001/archgenpsychiatry.2011.106. PMID 21969460
- [Background] Dawson G, Rogers S, Munson J, Smith M, Winter J, Greenson J, Donaldson A, Varley J. Randomized, controlled trial of an intervention for toddlers with autism: the Early Start Denver Model. Pediatrics. 2010 Jan;125(1):e17-23. doi: 10.1542/peds.2009-0958. Epub 2009 Nov 30. PMID 19948568
- [Background] Campbell DJ, Shic F, Macari S, Chawarska K. Gaze response to dyadic bids at 2 years related to outcomes at 3 years in autism spectrum disorders: a subtyping analysis. J Autism Dev Disord. 2014 Feb;44(2):431-42. doi: 10.1007/s10803-013-1885-9. PMID 23877749
- [Background] Farroni T, Csibra G, Simion F, Johnson MH. Eye contact detection in humans from birth. Proc Natl Acad Sci U S A. 2002 Jul 9;99(14):9602-5. doi: 10.1073/pnas.152159999. Epub 2002 Jun 24. PMID 12082186
- [Background] Kisilevsky BS, Hains SM, Brown CA, Lee CT, Cowperthwaite B, Stutzman SS, Swansburg ML, Lee K, Xie X, Huang H, Ye HH, Zhang K, Wang Z. Fetal sensitivity to properties of maternal speech and language. Infant Behav Dev. 2009 Jan;32(1):59-71. doi: 10.1016/j.infbeh.2008.10.002. Epub 2008 Dec 5. PMID 19058856
- [Background] Vouloumanos A, Hauser MD, Werker JF, Martin A. The tuning of human neonates' preference for speech. Child Dev. 2010 Mar-Apr;81(2):517-27. doi: 10.1111/j.1467-8624.2009.01412.x. PMID 20438457